CLINICAL TRIAL: NCT03750162
Title: Enterococcus Faecalis Elimination in Retreatment Cases Using Passive Ultrasonic Irrigation (PUI), Manual Dynamic Activation (MDA) and Photodynamic Therapy (PDT): a Randomized Clinical Trial
Brief Title: Bacteria Elimination in Retreatment Cases Using Different Disinfection Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Sevinç Aktemur Türker, Associate Professor, Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-27194235-02
Record Dates: First submitted 2018-11-18; First posted 2018-11-21 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Root Canal Infection; Periapical; Infection
Keywords: photodynamic therapy; diode laser
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Passive Ultrasonic irrigation (Experimental): Irrigation solution was ultrasonically activated in the canal for 1 minute by using IrriSafe tip coupled to an ultrasonic device with VDW Ultra .
  Interventions: Device: VDW Ultra
- Manuel dynamic activation (Experimental): Irrigation solution was activated with a well-fitting a ProtaperNext X3 gutta-percha point placed to working length was then moved in push - pull motions at a rate of 100 strokes/per minute
  Interventions: Device: ProtaperNext X3 gutta-percha
- Photodynamic Therapy (Experimental): Root canal was filled by 0.5 mL of 0.01% methylene blue (MB) solution for 5 minutes, then radiated by the light supply of a diode laser AMD picasso with a wavelength of 810 nm for 40 seconds (0.2 W).
  Interventions: Device: AMD picasso

INTERVENTIONS:
Device: VDW Ultra — supplementary disinfection technique
  Arms: Passive Ultrasonic irrigation
Device: AMD picasso — supplementary disinfection technique
  Arms: Photodynamic Therapy
Device: ProtaperNext X3 gutta-percha — supplementary disinfection technique
  Arms: Manuel dynamic activation

SUMMARY:
Nonsurgical root canal retreatment may become essential when the initial endodontic treatment fails because of the persistent intracanal or extracanal infections.It has been stated that the one of the main cause of posttreatment disease is the persistent or reintroduced microorganism such as enterococcus faecalis. Supplementary disinfection techniques such as irrigation agitation methods can help elimination of bacteria from root canal systems.

The aim of this in vivo study was to compare the effect of passive ultrasonic irrigation, manual dynamic activation and photodynamic therapy in reducing bacterial load in endodontic retreatment cases with periradicular lesion by using polymerase chain reaction (PCR)in a single visit root canal treatment.

DETAILED DESCRIPTION:
Thirty-six teeth with a single root and a single canal with posttreatment apical periodontitis which needed retreatment were selected for this study. Teeth were randomly divided into 3 groups according to the supplementary disinfection techniques used: Passive ultrasonic irrigation, Manual dynamic activation and Photodynamic therapy. Microbiological samples were taken before any intervention, after conventional chemo-mechanical preparation, and after disinfection techniques with sterile paper points and held in thioglycollate broth, and then were transferred to the microbiological laboratory. The amounts of e.faecalis in these samples was measured by using PCR.

ELIGIBILITY:
Inclusion Criteria:

Patients with no clinical symptoms Endodontically treated teeth Single rooted teeth

Exclusion Criteria:

Teeth with fractured instrument, resorption, perforation, ledge, over fillings Periodontal pockets deeper than 4 mm

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-09-05 (Actual)

PRIMARY OUTCOMES:
Bacteria change | 1 year
  Bacteria samples were taken at 3 step; before any intervention, after chemomechanical preparation, and after applying supplementary disinfection techniques

CONTACTS AND LOCATIONS:
Overall Officials: Sevinç Aktemur Türker, Study Director — Bulent Ecevit University
Locations (1):
- Bulent Ecevit University Faculty of Dentistry Department of Endodontics, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asnaashari M, Godiny M, Azari-Marhabi S, Tabatabaei FS, Barati M. Comparison of the Antibacterial Effect of 810 nm Diode Laser and Photodynamic Therapy in Reducing the Microbial Flora of Root Canal in Endodontic Retreatment in Patients With Periradicular Lesions. J Lasers Med Sci. 2016 Spring;7(2):99-104. doi: 10.15171/jlms.2016.17. Epub 2016 Mar 27. PMID 27330705
- [Background] Rodrigues RC, Antunes HS, Neves MA, Siqueira JF Jr, Rocas IN. Infection Control in Retreatment Cases: In Vivo Antibacterial Effects of 2 Instrumentation Systems. J Endod. 2015 Oct;41(10):1600-5. doi: 10.1016/j.joen.2015.06.005. Epub 2015 Jul 30. PMID 26234543